CLINICAL TRIAL: NCT06205771
Title: The Role and Mechanism of GPER Hippo Pathway in Regulating Uterine Arterial Smooth Muscle CBS/H2S in the Pathogenesis of Preeclampsia
Brief Title: The Role and Mechanism of GPER-Hippo-CBS/H2S Pathway in Preeclampsia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hao Feng (Other)
Responsible Party: Sponsor-Investigator, Hao Feng, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: YXLL-KY-2023（031）
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-01

CONDITIONS: Preeclampsia
Keywords: preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NP (No Intervention): normal pregnancy and preeclampsia pregnancy
- PE (Experimental): preeclampsia
  Interventions: Other: H2S content

INTERVENTIONS:
Other: H2S content — H2S content
  Arms: PE

SUMMARY:
The goal of this clinical trial is to learn about in health conditions. The main questions it aims to answer are:

* The pathological significance of GPER in uterine artery dilation in preeclampsia
* The Mechanism of GPER Hippo Pathway Regulating CBS/H2S in Human Uterine Artery Smooth Muscle Cells (hUASMC) This project intends to use GPER interfering RNA, YAP1 interfering RNA, in vivo perfusion experiments of human uterine artery tissue, and single cell patch clamp technology to study hypotheses under physiological/pathological pregnancy conditions at the tissue, cellular, and molecular levels, revealing a novel signal transduction pathway of estrogen stimulating vasodilation, providing new ideas for studying the mechanism of uterine artery blood flow regulation. This research result will provide new targets for intervention and treatment of diseases such as fetal intrauterine growth retardation and preeclampsia.

DETAILED DESCRIPTION:
1. Measure the content of H2S in uterine arterial smooth muscle and circulation of normal pregnancy and PE pregnant women, and analyze the relationship between the content of H2S in uterine arterial smooth muscle and circulation of PE pregnant women and PE.
2. Knock down the GPER and overexpression of GPER in HTR-8 cells, and detect the expression of GPER, CBS, and Hippo pathway related proteins using Western blot and qRT-PCR to verify the efficiency of knockdown and overexpression. Use different concentrations of H2S donor (GYY4137) to interfere with HTR-8 cells after treatment, and use RT-PCR and Western blot to detect the mRNA and protein expression of downstream molecules YAP and TAZ in Hippo pathway in cells, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Full term pregnancy with clinical diagnosis of preeclampsia and normal pregnancy pregnant woman
2. Pregnant women undergoing lower segment cesarean section for delivery

Exclusion Criteria:

1. Combined with chronic hypertension, kidney disease, intrahepatic cholestasis, etc Other basic diseases;
2. Multiple pregnancy
3. Pregnant women undergoing vaginal delivery
4. Normal pregnant women who are<37 weeks or>40 weeks pregnant

Max Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-04-10 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
H2S content in uterine arterial smooth muscle circulation | 8:00 am
  H2S content in circulation

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Shandong First Medical University &Shandong Provincial Qianfoshan Hospital, Jinan, Please Select, China

IPD SHARING:
Plan to Share IPD: Undecided